CLINICAL TRIAL: NCT06483776
Title: Kronik Obstrüktif Akciğer Hastalığında Düşmeye Etki Eden Faktörlerin Belirlenmesi
Brief Title: Determination of Factors Effecting Falls in Patients With COPD
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Principal investigator; PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: SBA 24/519
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Fall; Balance; Distorted
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD: Patients with Chronic Obstructive Pulmonary Disease

SUMMARY:
The aim of this study is to determine the factors affecting falls in patients with COPD.

DETAILED DESCRIPTION:
The aim of this study is to determine the factors affecting falls in patients with COPD. In accordance with the purposes, at least 100 patients with COPD who are 45-80 years old and clinically stable for four weeks will be included. Tests and questionnaires will be used in order to determine the severity of disease. Lung function test and respiratory muscle strength will be performed. Six Minute Walk Test and Six Minute Pegboard and Ring test will be performed with an armband that measures energy expenditure for functional exercise capacity for functional exercise capacity. To evaluate posture, the Corbin Postural Assessment Scale will be used. Hand grip test, periphreal muscle strength test, Time up and go test and One minute sit to stand test will be performed. International Physical Activity Questionnaire - Short Form (IPAQ) will be used to determine physical activity level. Mini- Besttest and Activity-specific Balance Confidence Scale were used to determine fall risk. According to the results to be obtained factors affecting falls will be determined in patients with COPD. It will guide professional working in this field.

ELIGIBILITY:
Inclusion Criteria for Chronic Obstructive Pulmonary Disease Group;

* Being between the ages of 45 and 80,
* Being literate,
* Willing to participate in the study,
* Having COPD classified as stage 1-2-3-4 according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) system,
* Being clinically stable for the past 4 weeks.

Exclusion Criteria for Chronic Obstructive Pulmonary Disease Group;

* Having a history of lung cancer, sarcoidosis, tuberculosis, and/or lung surgery,
* Having any neurological, neuromuscular, vestibular, or cardiac disease that could affect the measurements,
* Receiving long-term oxygen therapy.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD s will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Balance and Fall risk | 1 day
  Time up and go test will be used to assess balance and fall risk. The cut off point will be determined as 12 second for patients with COPD.
Balance and Fall risk-The Mini-Balance Evaluation Systems Test (Mini-BESTest) | 1 day
  It will be used to evaluate individuals' static and dynamic balance. It consists of four sub-parameters: preparatory movements, reactive postural control, sensory orientation, and dynamic gait, with a total of four items. The test, which takes an average of 10-15 minutes to complete, is evaluated out of a total of 28 points. A higher score indicates higher function. This test is valid and reliable in patients with COPD.
Balance and Fall risk- The Activities-specific Balance Confidence scale (ABC scale) | 1 day
  It will be used to evaluate fall risk. A validity and reliability study has been conducted in Turkish. This scale assesses balance confidence based on functional status with 16 task-specific questions. Each question is scored between 0% (no confidence) and 100% (full confidence), and a higher total score indicates higher confidence. Scores below 67% indicate fall risk in elderly individuals. It is valid and reliable for determining fall risk in individuals with COPD.

SECONDARY OUTCOMES:
Functional exercise capacity | 1 day
  Functional exercise capacity will be determined via Six Minute Walk Test.
Respiratory Muscle Strength | 1 day
  Respiratory muscle strength will be assessed via a using a mouth pressure device according to American Thoracic Society/ European Respiratory Society guidelines.
Posture | 1 day
  Posture will be examined via the Corbin Postural Assessment Scale. The total points of the Corbin Postural Assessment Scale range from 0 to 28 points. A higher point represents worse posture.
Dyspnea | 1 day
  The Modified Medical Research Council will be used for patients with COPD. The Modified Medical Research Council consist of five grades. A higher grades represents severe dyspnea level.
Symptoms | 1 day
  Chronic Obstructive Pulmonary Disease Assessment Test will be used to determine symptoms. The total score of Chronic Obstructive Pulmonary Disease Assessment Test changes from 0 to 40 points, and 10 points is the accepted cut-off point for COPD.
Severity of disease | 1 day
  Global Initiative for Chronic Obstructive Pulmonary Disease and Global Initiative for Chronic Obstructive Pulmonary ABE assessment Tool will be used for severity of disease. According to the Global Initiative for Chronic Obstructive Pulmonary Disease, the severity of airflow limitation (Forced Expiratory Volume in 1 s) was determined as mild (≥ 80%), moderate (50-80%), severe (30-50%), and very severe (<30%). According to Global Initiative for Chronic Obstructive Pulmonary A,B,E assessment Tool, patients classified group A, B, and E using symptom status and airflow limitation.
Peripheral muscle strength | 1 day
  Peripheral muscle strength will be assessed via hand dynamometer.
Lower extremity capacity | 1 day
  One minute sit to stand test will be used for lower extremity capacity.
Hand grip test | 1 day
  Hand grip will be evaluated via hand dynamometer.
Energy expenditure | 1 day
  An armband will be used to assess energy expenditure during six minute walk test and six minute pegboard and ring test.
Physical activity | 1 day
  Individuals' physical activity levels will be assessed using the International Physical Activity Questionnaire - Short Form. The questionnaire, developed by Craig et al. (2003), has been validated and tested for reliability in Turkish by Öztürk et al. (2005). In the assessment of activities, each activity must be performed for at least 10 minutes at a time. The IPAQ short form provides information about time spent sitting, walking, in moderate-intensity activities, and in vigorous-intensity activities. A score is obtained by multiplying the duration in minutes, the number of days, and the MET (metabolic equivalent) value, resulting in a "MET-minutes/week" score. According to the scoring system, the intensity of physical activity is classified as low if the score is less than 600 MET-minutes/week, moderate if between 600 and 3000, and high if more than 3000.
Upper Extremity Functional Capacity | 1 day
  Upper extremity functional capacity will be assessed by six minute pegboard and ring test in patients with COPD
Bode index | 1 day
  It will be used to assess the risk of mortality due to COPD. This assessment includes body mass index (BMI), airway obstruction (FEV1 % predicted), dyspnea (mMRC dyspnea score), and exercise capacity (6-minute walk distance) in this index. BMI >21 is scored as 0, and ≤21 is scored as 1. Airway obstruction reflected by FEV1 (% predicted) is scored as follows: ≥65 is 0, 50-64 is 1, 36-49 is 2, and ≤35 is 3. The degree of dyspnea according to the mMRC scale is scored as follows: mMRC scores 0-1 are 0 in the BODE index, 2 is 1, 3 is 2, and 4 is 3. Finally, for exercise capacity, a 6MWD ≥350m is scored as 0, 250-349m is 1, 150-249m is 2, and ≤149m is 3 in the BODE index. The total score is determined by summing the individual scores. The BODE index can predict not only mortality but also the risk of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PT, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)